CLINICAL TRIAL: NCT00983294
Title: A One-Directional, Open-Label Drug Interaction Study to Investigate the Effects of Multiple-Dose Azithromycin on Single-Dose Pharmacokinetics of Colchicine in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study of Colchicine and Azithromycin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mutual Pharmaceutical Company, Inc. (Industry)
Responsible Party: Vice President, Branded Products and Medical Affairs, Mutual Pharmaceutical Company, Inc.
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MPC-004-08-1011
Record Dates: First submitted 2009-08-13; First posted 2009-09-24 (Estimated); Results first posted 2009-09-24 (Estimated); Last update posted 2009-10-28 (Estimated); Status verified 2009-10

CONDITIONS: Pharmacokinetics
Keywords: blood levels over time;; colchicine;; azithromycin;; healthy
MeSH Terms: interventions — Colchicine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colchicine alone (Active Comparator): baseline colchicine pharmacokinetics
  Interventions: Drug: Colchicine
- Colchicine with steady-state Azithromycin (Experimental): colchicine pharmacokinetics in presence of steady-state azithromycin
  Interventions: Drug: Azithromycin; Drug: Colchicine

INTERVENTIONS:
Drug: Colchicine — A single dose of 0.6 mg colchicine administered alone at 7:30 am on Day 1
  Other Names: COLCRYS™
  Arms: Colchicine alone
Drug: Azithromycin — Two 250 mg azithromycin tablets administered at 7:30 am on Day 15, then one 250 mg tablet administered daily at 7:30 am on Days 16 to 19.
  Other Names: Zithromax® Tablets USP, 250 mg
  Arms: Colchicine with steady-state Azithromycin
Drug: Colchicine — A single dose of 0.6 mg colchicine administered with azithromycin at 7:30 am on Day 19.
  Other Names: COLCRYS™
  Arms: Colchicine with steady-state Azithromycin

SUMMARY:
Azithromycin is a possible weak to moderate inhibitor of CYP3A4, one of the enzymes responsible for the metabolism of colchicine. This study will evaluate the effect of multiple doses of azithromycin on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. A secondary objective is to evaluate the safety and tolerability of this regimen in healthy volunteers. All study subjects will be monitored for adverse events throughout the study period.

DETAILED DESCRIPTION:
Azithromycin is a possible weak to moderate inhibitor of CYP3A4, one of the enzymes responsible for the metabolism of colchicine. This study will evaluate the effect of multiple doses of azithromycin on the pharmacokinetic profile of a single 0.6 mg dose of colchicine. On day 1, after a fast of at least 10 hours, twenty-four healthy non-smoking, non-obese, non-pregnant adult volunteers between the ages of 18 and 45 will be given a single oral dose of colchicine 0.6 mg. Fasting will continue for 4 hours after the dose. Blood samples will be drawn from all participants before dosing and for twenty-four hours post-dose on a confined basis at times sufficient to adequately define the pharmacokinetics of colchicine. Blood sampling will then continue on a non-confined basis on Days 2-5. After a 2 week washout period, beginning on Day 15 and continuing through day 18, subjects will return to the clinic daily for non-confined dosing of azithromycin given orally 2 x 250 mg tablets on Day 15 followed by 1 x 250 mg tablet on Days 16-18. Administered azithromycin doses on these days will not necessarily be in a fasted state. On Day 15 after taking the first dose of azithromycin, subjects will remain in the clinic for observation for 1 hour post-dose administration. On Day 19, after a fast of at least 10 hours, all study subjects will receive a co-administered single dose of colchicine (0.6 mg) and azithromycin (1 x 250 mg tablet). All subjects will be confined to the clinic for the 24-hour period following the dose. Blood will be drawn at time sufficient to define the pharmacokinetics of colchicine in the presence of azithromycin at steady state. Blood sampling will continue on a non-confined basis on Days 20-23. A further goal of this study is to evaluate the safety and tolerability of this regimen in healthy volunteers. Subjects will be monitored throughout participation in the study for adverse reactions to the study drug and/or procedures. Seated blood pressure and pulse will be measured prior to dosing and at approximately 1, 2, and 3 hours following drug administration on Days 1 and 19. All adverse events whether elicited by query, spontaneously reported, or observed by clinic staff will be evaluated by the Investigator and reported in the subject's case report form.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-45 years of age, non-smoking and non-pregnant (postmenopausal, surgically sterile or using effective contraceptive measures) with a body mass index (BMI) greater than or equal to 18 and less than or equal to 32, inclusive

Exclusion Criteria:

* Recent participation (within 28 days) in other research studies
* Recent significant blood donation
* Pregnant or lactating
* Test positive at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV)
* Recent (2-year) history or evidence of alcoholism or drug abuse
* History or presence of significant cardiovascular, pulmonary, hepatic, gall bladder or biliary tract, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease Subjects who have used any drugs or substances known to inhibit or induce cytochrome (CYP) P450 enzymes and/or P-glycoprotein (P-gp) within 28 days prior to the first dose and throughout the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony R Godfrey, Pharm.D., Principal Investigator — PRACS - Cetero

REFERENCES:
- [Derived] Terkeltaub RA, Furst DE, Digiacinto JL, Kook KA, Davis MW. Novel evidence-based colchicine dose-reduction algorithm to predict and prevent colchicine toxicity in the presence of cytochrome P450 3A4/P-glycoprotein inhibitors. Arthritis Rheum. 2011 Aug;63(8):2226-37. doi: 10.1002/art.30389. PMID 21480191
- See also: Recalls, Market Withdrawals and Safety Alerts — http://www.fda.gov/opacom/7alerts.html
- See also: Daily Med - Posting of Recently Submitted Labeling to the FDA — http://dailymed.nlm.nih.gov/dailymed/about.cfm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-four (24) healthy, non-smoking, male and female volunteers, consisting of members of the community at large, were to be enrolled.
Pre-assignment Details: 40 subjects screened, 6 were screen failures, 6 had schedule conflicts, 3 transferred to another study, 1 was not needed
Groups:
- Colchicine Alone / With Azithromycin (at Steady State): [All subjects received each of the study treatments.] Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:30 am after an overnight fast, followed by a washout period of 14 days. On Day 15, each subject received two 250 mg azithromycin tablets at 7:30 am after an overnight fast, followed by one 250 mg azithromycin tablet daily at 7:30 am without regard to meals on Days 16 to 18. Then, on Day 19, each subject received both one 0.6 mg colchicine tablet and one 250mg azithromycin tablet at 7:30 am after an overnight fast.
Period: Colchicine Alone
Arm/Group | Colchicine Alone / With Azithromycin (at Steady State)
Started | 24
Completed | 24
Not Completed | 0
Period: 14 Day Washout Period
Arm/Group | Colchicine Alone / With Azithromycin (at Steady State)
Started | 24
Completed | 22 (two subjects withdrew consent due to personal reasons)
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Azithromycin Alone
Arm/Group | Colchicine Alone / With Azithromycin (at Steady State)
Started | 22
Completed | 22
Not Completed | 0
Period: Colchicine With Azithromycin
Arm/Group | Colchicine Alone / With Azithromycin (at Steady State)
Started | 22
Completed | 21 (withdrawn by sponsor on Day 21 due to vomiting on Day 15, prior to azithromycin dosing(1))
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Colchicine Alone / With Azithromycin (at Steady State): [All subjects received each of the study treatments.] Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:30am after an overnight fast, followed by a washout period of 14 days. On Day 15, each subject received two 250 mg azithromycin tablets at 7:30 am after an overnight fast, followed by one 250 mg azithromycin tablet daily at 7:30 am without regard to meals on Days 16 to 18. Then, on Day 19, each subject received both one 0.6 mg colchicine tablet and one 250 mg azithromycin tablet at 7:30 am after an overnight fast.
Arm/Group | Colchicine Alone / With Azithromycin (at Steady State)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants] — age range: >=18 and <=45
  Participants
    <=18 years | 0
    Between 18 and 65 years | 24
    >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 27.7 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: The maximum or peak concentration that colchicine reaches in the plasma.
Time Frame: serial pharmacokinetic plasma concentrations were drawn prior to colchicine dose administration (0 hour) on Days 1 and 19, then at 0.5, 1.0, 1.5, 2, 3, 4, 5, 6, 8, 12, 24, 36, 48, 72, and 96 hours after colchicine dose administration
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Colchicine Alone: On Day 1, each subject received one 0.6 mg colchicine tablet at 7:30 am after an overnight fast, followed by a washout period of 14 days.
- Colchicine With Azithromycin (at Steady-state): On Day 15, each subject received two 250 mg azithromycin tablets at 7:30 am after an overnight fast, followed by one 250 mg azithromycin tablet daily at 7:30 am without regard to meals on Days 16 to 18. Then, on Day 19, each subject received both one 0.6 mg colchicine tablet and one 250 mg azithromycin tablet at 7:30 am after an overnight fast.
Arm/Group | Colchicine Alone | Colchicine With Azithromycin (at Steady-state)
Number analyzed (Participants) | 21 | 21
pg/mL | 2,737.00 (1,136.28) | 3,051.76 (1,206.72)

2. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 to Time t [AUC(0-t)]
Description: The area under the colchicine plasma concentration versus time curve, from time 0 to the time of the last measurable colchicine concentration (t), as calculated by the linear trapezoidal rule.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Azithromycin (at Steady-state)
Number analyzed (Participants) | 21 | 21
pg-hr/mL | 11,975.72 (5,485.83) | 17,161.00 (6,482.74)

3. Primary Outcome: Area Under the Concentration Versus Time Curve From Time 0 Extrapolated to Infinity [AUC(0-∞)]
Description: The area under the colchicine plasma concentration versus time curve from time 0 to infinity. AUC(0-∞) was calculated as the sum of AUC(0-t) plus the ratio of the last measurable colchicine plasma concentration to the elimination rate constant.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg-hr/mL
Arm/Group | Colchicine Alone | Colchicine With Azithromycin (at Steady-state)
Number analyzed (Participants) | 21 | 21
pg-hr/mL | 14,125.25 (6,600.26) | 19,611.01 (7,678.56)

ADVERSE EVENTS:
Groups:
- Colchicine Alone: Each subject received one 0.6 mg colchicine tablet on Day 1 at 7:30am after an overnight fast, followed by a washout period of 14 days.
- Azithromycin Alone: On Day 15, each subject received two 250mg azithromycin tablets at 7:30 am after an overnight fast, followed by one 250mg azithromycin tablet daily at 07:30 without regard to meals on Days 16 to 18.
- Colchicine With Steady-state Azithromycin: On Day 19, each subject received both one 0.6mg colchicine tablet and one 250mg azithromycin tablet at 07:30 after an overnight fast.
Arm/Group | Colchicine Alone | Azithromycin Alone | Colchicine With Steady-state Azithromycin
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 8 | 5 | 4
OTHER ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Colchicine Alone | Azithromycin Alone | Colchicine With Steady-state Azithromycin
cardiac flutter (Cardiac disorders) | 0/24 (0) | 0/22 (0) | 1/22 (1)
palpitations (Cardiac disorders) | 1/24 (1) | 0/22 (0) | 1/22 (1)
abdominal pain upper (Gastrointestinal disorders) | 0/24 (0) | 2/22 (2) | 1/22 (1)
diarrhoea (Gastrointestinal disorders) | 2/24 (2) | 0/22 (0) | 0/22 (0)
nausea (Gastrointestinal disorders) | 0/24 (0) | 0/22 (0) | 2/22 (3)
stomach discomfort (Gastrointestinal disorders) | 1/24 (1) | 0/22 (0) | 0/22 (0)
vomiting (Gastrointestinal disorders) | 1/24 (1) | 1/22 (1) | 0/22 (0)
back pain (Musculoskeletal and connective tissue disorders) | 1/24 (1) | 0/22 (0) | 0/22 (0)
musculoskeletal stiffness (Gastrointestinal disorders) | 1/24 (1) | 0/22 (0) | 0/22 (0)
dizziness (Nervous system disorders) | 1/24 (1) | 0/22 (0) | 0/22 (0)
headache (Nervous system disorders) | 3/24 (4) | 2/22 (2) | 1/22 (1)
paraesthesia (Nervous system disorders) | 0/24 (0) | 0/22 (0) | 1/22 (1)
somnolence (Nervous system disorders) | 0/24 (0) | 1/22 (1) | 0/22 (0)
syncope (Nervous system disorders) | 1/24 (1) | 0/22 (0) | 0/22 (0)
insomnia (Psychiatric disorders) | 1/24 (1) | 0/22 (0) | 0/22 (0)
pollakiuria (Renal and urinary disorders) | 1/24 (1) | 0/22 (0) | 0/22 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days